CLINICAL TRIAL: NCT00580411
Title: A Timeline Study of Alcohol Use and Its Relationship to Insomnia
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Principal Investigator, Principal Investigator, National Institute on Drug Abuse (NIDA)
Other Study IDs: HR#16934; Contract ID ESRC343; DPMCDA
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2015-10

CONDITIONS: Insomnia; Alcohol Problem
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alcohol-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alcohol Problem First: Alcohol Problem precedes Insomnia
- Insomnia First: Insomnia Precedes Alcohol Problem

SUMMARY:
This study is an epidemiological and descriptive study of the lifetime relationship of insomnia to alcohol problems.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages of 18-70, may be male or female, and from any ethnic background.
* Individuals must have the capacity to give IRB-approved study consent.
* Subjects must at least have a lifetime history of being heavy alcohol drinkers (i.e., drinks approximately 21 alcoholic drinks or more per week). Alternatively, subjects are eligible if they meet criteria for a lifetime history of either alcohol dependence or alcohol abuse. Overall, a subject must meet at least one of these alcohol criteria: a lifetime history of heavy drinking, alcohol abuse or alcohol dependence.
* Subjects must have a complaint of chronic insomnia, reporting either six or less hours TST, on average at least three times per week.

Exclusion Criteria

* Potential subjects with a lifetime diagnosis of Bipolar Affective Disorder, Schizophrenia, Borderline Personality Disorder, dementia of any type, or epilepsy will not be admitted to the study.
* Subjects will be excluded with a diagnosis of any other substance dependence syndrome other than alcohol dependence, nicotine dependence, and/or caffeine dependence. However, individuals may have a history of episodic abuse of cannabis, cocaine, sedatives/hypnotics and opiates, amphetamines, and hallucinogens. Also, subjects may be on prescription benzodiazepine or related sedative/hypnotic therapy.
* Any condition or treatment of a condition that is likely to confound the experimental design or the results will be prohibited by the PI.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We wish to study individuals who meet lifetime criteria for alcohol dependence, abuse or heavy drinking and who self-report current insomnia.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2007-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To characterize the temporal relationship between insomnia and alcohol dependence, alcohol abuse or heavy drinking and determine if this relationship affects the severity of alcohol use. | Visit 1

SECONDARY OUTCOMES:
To assess the utility of 3 sleep disorder instruments: the ISI, the SDQ-8 & the ESS in an inpatient or outpatient population of subjects reporting insomnia with a lifetime history of alcohol dependence, alcohol abuse or heavy drinking. | Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Robert Malcolm, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States